CLINICAL TRIAL: NCT03990818
Title: Continuous Registration of Bioimpedance During Hemodialysis
Acronym: DELAGE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mode Sensors AS (Industry)
Collaborators: Helse Nord-Trøndelag HF (Other)
Responsible Party: Sponsor
Other Study IDs: 2019 DELAGE
Record Dates: First submitted 2019-06-17; First posted 2019-06-19 (Actual); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: Dialysis Related Complication; Dehydration
MeSH Terms: conditions — Dehydration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This studies aims at testing continuous registration of bioimpedance during hemodialysis and comparing the measurement with extracted liquid.

DETAILED DESCRIPTION:
The purpose is to test the sensitivity and specificity of a new electronic patch in the indication of the relative change in the fluid balance. If possible, the change in hydration level should be quantified. The test is done on patients during hemodialysis. Extracted amount of fluid is used as the primary reference to the bioimpedance measurements, but other references will also be used.

The measurement is made using bioimpedance measured with four electrodes and over a large frequency spectrum. Impedance measurements are made every 20 seconds throughout the test period. The measurement is recorded in a memory (flash) on each patch. At the same time as measuring bioimpedance, the temperature in the patch is recorded.

After completion of the test, the data is transferred to a computer for analysis. As a reference, extracted amount of fluid, weight change, blood samples and clinical evaluation are used.

ELIGIBILITY:
Inclusion Criteria:

* Patients for hemodialysis

Exclusion Criteria:

* Acute in-current disease.
* Known adverse reaction to medical adhesive

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients for hemodialysis
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2019-08-20 (Actual); Primary Completion 2019-09-30 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of patch performance | August - December 2019
  Establish sensitivity and specificity of patch performance relative to extracted water, weight change and blood sample results

CONTACTS AND LOCATIONS:
Overall Officials: Magnus Nordahl, Study Chair — Mode Sensors AS
Locations (1):
- Levanger Hospital, Levanger, Norway